CLINICAL TRIAL: NCT06364748
Title: Expanding Access to Care Through Telemedical Support for Vital Sign Monitoring in High-risk Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Michigan Cancer Center (Other)
Collaborators: Veta Health (Unknown)
Responsible Party: Principal Investigator, David Shalowitz, Principal Investigator, West Michigan Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 002-2024-Shalowitz
Record Dates: First submitted 2024-03-05; First posted 2024-04-15 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Smart Cuff Group (Active Comparator): Smart blood pressure cuff
  Interventions: Device: Cellular enabled blood pressure cuff
- Control Group (Placebo Comparator): Standard of care
  Interventions: Device: Standard of Care Cuff

INTERVENTIONS:
Device: Cellular enabled blood pressure cuff — Smart cuff
  Arms: Smart Cuff Group
Device: Standard of Care Cuff — Standard blood pressure cuff
  Arms: Control Group

SUMMARY:
A randomized trial of remote blood pressure monitoring, compared to usual care, in patients receiving bevacizumab to determine whether remote blood pressure monitoring improves the collection of blood pressure data, identification and management of clinically significant hypertension, and patient satisfaction.

DETAILED DESCRIPTION:
Remote patient monitoring (RPM) technology has the potential to improve the early detection and management of clinically significant hypertension in cancer patients undergoing therapy with bevacizumab, by allowing immediate communication of abnormal measurements to the clinical care team. Additionally, RPM may decrease patients' and caregivers' burdens of ongoing cancer care through an improved user experience compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a male or female 18 years of age or older.
2. Participant is a current patient at West Michigan Cancer Center/Bronson Cancer Center.
3. Participant is receiving bevacizumab as part of active treatment.
4. Participant is willing and able to provide written informed consent.

Exclusion Criteria:

1. Participant is unable to understand English.
2. Participant is hospitalized.
3. Participants are unable to obtain blood pressure readings at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
To determine whether remote blood pressure monitoring improves adherence to recommendations for daily systolic and diastolic blood pressure monitoring compared to usual care | Through study completion, an average of 12 weeks
  Comparing the number of participants who complete the recommended daily blood pressure readings available for clinician assessment via review of a remote blood pressure monitoring platform versus a patient recorded blood pressure log book

SECONDARY OUTCOMES:
Improvement of early identification of bevacizumab-induced hypertension with usual care blood pressure monitoring | Through study completion, an average of 18 months
  Frequency of clinician notifications of clinically significant elevations in systolic and/or diastolic blood pressure readings
Improvement of early identification of bevacizumab-induced hypertension with remote blood pressure monitoring | Through study completion, an average of 18 months
  Frequency of clinician notifications of clinically significant elevations in systolic and/or diastolic blood pressure readings
Patient satisfaction with usual care blood pressure monitoring | 1 week after enrollment, 6 weeks after enrollment and 12 weeks after enrollment
  Patient questionnaire containing seven questions, using a 5-point Likert scale, where 1 equals "Strongly Disagree" and 5 equals "Strongly Agree" for six questions. One question is measured using a 5-point Likert scale, where 1 equals "Very Difficult" and five equals "Not Difficult At All"
Patient satisfaction with remote blood pressure monitoring | 1 week after enrollment, 6 weeks after enrollment and 12 weeks after enrollment
  Patient questionnaire sent via mobile application by Veta Health, containing seven questions, using a 5-point Likert scale, where 1 equals "Strongly Disagree" and 5 equals "Strongly Agree" for six questions. One question is measured using a 5-point Likert scale, where 1 equals "Very Difficult" and five equals "Not Difficult At All"

CONTACTS AND LOCATIONS:
Overall Officials: David Shalowitz, Principal Investigator — West Michigan Cancer Center
Locations (1):
- West Michigan Cancer Center, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No